CLINICAL TRIAL: NCT06376799
Title: Which Health-care Professional(s) to Talk About Advance Care Planning ? The Point of View of French Patients Followed in the Context of an Oncological Disease.
Brief Title: Which Health-care Professional(s) to Talk About Advance Care Planning ?
Acronym: QPSPAS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC23.0437; 2024-A00485-42 (Other: ID RCB)
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Advance Care Planning; Patient Preference
Keywords: Advance care planning; Patient preference
MeSH Terms: conditions — Patient Preference

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- French adult patients followed in the context of a oncological disease,: French-speaking adult patients willing to participate in this study. Patients being treated for oncological disease, in a curative, palliative, or remission phase.
  Interventions: Other: Self-questionnaire

INTERVENTIONS:
Other: Self-questionnaire — Provision of a self-questionnaire in digital or paper format for the patient. The patient will be asked to indicate their preferences regarding the primary and secondary objectives of the study.

SUMMARY:
The goal of this descriptive observational study is to evaluate the preference of French adult patients followed in the context of a oncological disease, regarding the choice of the preferred healthcare professional to discuss advance care planning.

To this end, voluntary participants will be asked to indicate their preferences by answering a self-questionnaire available in electronic or paper format.

ELIGIBILITY:
Inclusion Criteria :

* Patients with neoplasic disease (under treatment, in exclusive palliative phase, under surveillance or in remission)
* French-speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The source population corresponds to the French-speaking population of the Grenoble metropole area, followed in the context of cancer and treated by community medicine and/or healthcare structures.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-02 (Estimated)

PRIMARY OUTCOMES:
Determining the healthcare professional preferred by cancer patients to talk about advance care planning | Six months
  Hierarchical classification of healthcare professionals preferred by the patient via a self-questionnaire

SECONDARY OUTCOMES:
Determining cancer patients' second choice of healthcare professional to talk about advance care planning | Six months
  Hierarchical classification of health professionals preferred as second choice via a self-questionnaire
Evaluation of patient preferences regarding advance care planning, concerning the form, the moment it should be carried out, whether or not they wish to be accompanied by a relative, and the benefit of systematization | Six months
  Percentage for each response to the questions relating to the modalities of carrying out the interview regarding advance care planning; the most relevant time to discuss advance care planning; the patient's wish to be accompanied or not by a relative at the time of this interview; and the patient's opinion on the relevance of systematically carrying out this interview.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rietjens JAC, Sudore RL, Connolly M, van Delden JJ, Drickamer MA, Droger M, van der Heide A, Heyland DK, Houttekier D, Janssen DJA, Orsi L, Payne S, Seymour J, Jox RJ, Korfage IJ; European Association for Palliative Care. Definition and recommendations for advance care planning: an international consensus supported by the European Association for Palliative Care. Lancet Oncol. 2017 Sep;18(9):e543-e551. doi: 10.1016/S1470-2045(17)30582-X. PMID 28884703
- [Background] Brinkman-Stoppelenburg A, Rietjens JA, van der Heide A. The effects of advance care planning on end-of-life care: a systematic review. Palliat Med. 2014 Sep;28(8):1000-25. doi: 10.1177/0269216314526272. Epub 2014 Mar 20. PMID 24651708
- [Background] Peck V, Valiani S, Tanuseputro P, Mulpuru S, Kyeremanteng K, Fitzgibbon E, Forster A, Kobewka D. Advance care planning after hospital discharge: qualitative analysis of facilitators and barriers from patient interviews. BMC Palliat Care. 2018 Dec 5;17(1):127. doi: 10.1186/s12904-018-0379-0. PMID 30518345
- [Background] Kubi B, Istl AC, Lee KT, Conca-Cheng A, Johnston FM. Advance Care Planning in Cancer: Patient Preferences for Personnel and Timing. JCO Oncol Pract. 2020 Sep;16(9):e875-e883. doi: 10.1200/JOP.19.00367. Epub 2020 Apr 13. PMID 32282265